CLINICAL TRIAL: NCT02795884
Title: Adjuvant Erlotinib Intercalating Chemotherapy or Adjuvant Chemotherapy Alone in NSCLC With Common EGFR Mutation
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of reconsideration of using erlotinib(EGFR Tyrosine kinase inhibitor) as adjuvant aim
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0926
Record Dates: First submitted 2016-02-24; First posted 2016-06-10 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: NSCLC
Keywords: Lung cancer; NSCLC; adjuvant treatment
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Erlotinib Hydrochloride; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intercalation arm (Experimental): * Intercalation phase (Duration: 3wks x 4 cycles = 12 wks) Pemetrexed 500mg/m2 D1, Cisplatin 75mg/m2 D1, Erlotinib 150mg D8-21 q3wks
  * Maintenance phase (Duration: 1 year) Erlotinib 150mg D1-28
  Interventions: Drug: intercalation therapy using pemetrexed, cisplatin and erlotinib
- Chemotherapy alone arm (Active Comparator): Duration: 3wks x 4 cycles = 12 wks Vinorelbine 25mg/m2 D1,8, Cisplatin 75mg/m2 D1 q3wks
  Interventions: Drug: Vinorelbine, cisplatin

INTERVENTIONS:
Drug: intercalation therapy using pemetrexed, cisplatin and erlotinib — During the intercalation phase of the initial 12-week period, erlotinib is to be orally administered at the dose of 150 mg daily from Day 8 to Day 21 at every cycle of 21 days. During the maintenance phase after 12 weeks, it is orally administered at the cycle of 28 days without a wash-out period at the dose of 150 mg daily for one year. The combination of pemetrexed and cisplatin will be administered for 4 cycles in total by each cycle of 21 days, and it is to be administered by intravenous (IV) infusion on every Day 1. Pemetrexed 500 mg/m2 will be diluted in 100 ml of 0.9% saline solution and will be administered by intravenous (IV) infusion for 10 minutes. Cisplatin 75 mg/m2 will be diluted in 150 ml of 0.9% saline solution and will be administered by intravenous (IV) infusion for 10 to 15 minutes. The combination of pemetrexed and cisplatin will be administered for 4 cycles in total by each cycle of 21 days, and it is to be administered by intravenous (IV) infusion on every Day 1.
  Arms: Intercalation arm
Drug: Vinorelbine, cisplatin — Vinorelbine 25mg/m2 will be diluted in 50 ml of 0.9% saline solution and will be administered by intravenous (IV) infusion for 6 to 10 minutes and then wash the catheter using 100 ml of 0.9% saline solution. Cisplatin 75 mg/m2 will be diluted in 150 ml of 0.9% saline solution and will be administered by intravenous (IV) infusion for 10 to 15 minutes.
  Arms: Chemotherapy alone arm

SUMMARY:
This study will be performed as a local multicenter, randomized, phase III clinical study. It will compare the adjuvant chemotherapy in Stage IB-IIIA NSCLC with common EGFR mutation (Exon 19 deletion or L858R) who underwent total resection and the Erlotinib-Intercalation adjuvant chemotherapy with the chemotherapy alone. The patients will be randomly assigned to the Intercalation combination chemotherapy regimen and the chemotherapy alone regimen at the ratio of 1:1. The treatment regimen of each arm is as follows.

ELIGIBILITY:
Inclusion Criteria:

* A screening examination should be implemented within 14 after obtaining the informed consent, and the treatment should be started within 14 days after the randomization of subjects. Subjects who are applicable to all of the following criteria will be eligible for inclusion in this clinical study.

  * Stage IB-IIIA Non-squamous NSCLC (Based on AJCC Version 7 TNM Disease Stages)
  * Surgically complete resection
  * Confirmed with Exon 19 deletion or L858R EGFR mutation
  * Complete recovery from the surgery. The period up to the post-operative randomization can be 3 weeks at minimum up to 8 weeks at maximum.
  * Age to be ≥ 19 years old
  * Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
  * Patients who are not pregnant or breastfeeding
  * Appropriate functions of bone marrow, liver and kidney, when assessed with the following requirements of the laboratory tests to be conducted within 14 days before the initial dose of the study drug:
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 times greater than the upper limit of normal
  * ALT and AST ≤ 2.5 times greater than the upper limit of normal
  * Alkaline phosphatase ≤ 2.5 times greater than the upper limit of normal
  * INR and PTT ≤ 1.5 times greater than the upper limit of normal
  * Appropriate renal function: Serum creatinine ≤ 1.25 × upper limit of normal, or serum creatinine clearance according to Cockcroft-Gault formula(below) ≥50 mL/min

Woman CrCl = (140- age [years old]) x weight (kg) x 0.85 72 x serum creatinine (mg/dL)

Man CrCl = (140- age [years old]) x weight (kg) x 1.00 72 x serum creatinine (mg/dL)

* Patients who are capable of complying with the clinical study protocol and who can take medication orally
* Patient who can hear sufficient explanation and sign on the informed consent form

Exclusion Criteria:

* Any subject who shows any of the following criteria should be excluded from this clinical study:

  * Patient identified with T790M mutation
  * Treatable with topical treatments (radiotherapy or surgery)
  * Previous treatment to inhibit the human epidermal growth factor receptor (EGFR) (e.g. erlotinib, gefitinib, cetuximab, trastuzumab, etc.)
  * Prior systemic chemotherapy
  * Any prior known hypersensitive reaction to the study agents
  * CTCAE> grade 2 clinically significant active infection
  * Any known infection with Human Immunodeficiency Virus (HIV) or chronic hepatitis type B or type C virus For the patients positive to chronic hepatitis type B or type C virus without elevation of AST/ALT, their inclusion/exclusion will be determined at the discretion of the investigator.
  * Seizures in need of treatment (steroid or antiepileptic treatment)
  * Medical history of interstitial lung disease
  * Medical history of organ allograft within six months
  * Subjects under dialysis
  * A subject diagnosed with another cancer within 3 years before participating in this clinical study (treated carcinoma in situ of the cervix, treated skin basal cell carcinoma, and treated superficial bladder tumors [Ta and Tis] will not be applicable). For surgically completely resected thyroid cancer, it will be determined at the discretion of the investigator.
  * Unstable or any status that would potentially put the subject in danger or that would interfere with compliance of the subject in the clinical study.
  * Treatment with the investigational products other than the one to be used in this clinical study during participation in the clinical study or within 4 weeks prior to participation in the clinical study
  * Pregnant or breastfeeding women. The women at childbearing ages should show negative response to the serum pregnancy test being conducted within 7 days before the initial administration of the study drug. Not only the women at childbearing ages, but also men who give consent to use appropriate contraceptive methods before entering the clinical study and during the period of the clinical study including 30 days after the last dose of the study drug. Post-menopausal women are defined as:

    1. With no menstruation at least for 12 months, at the age >50 years old, or
    2. With no natural menstruation at least for 6 months and the level of follicle-stimulating hormone (FSH) is in the post-menopausal range (>40 mIU/mL) at the age ≤50 years old, or
    3. Bilateral oophorectomy Men and women who are to be enrolled in this clinical study must use appropriate blocking contraceptive methods in prior to and during the clinical study. Appropriate contraceptive methods include implant or combined oral contraceptive agent-utilized hormone contraception, some intrauterine contraceptive device, bilateral tubal ligation, hysterectomy, or vasectomy of the partner. In addition, use of condom is required for the subject or his/her partner.
  * Subjects who are unable to swallow oral medication or with all types of absorption disorders
  * In addition, when the investigator determines it is not adequate to perform the study due to serious systemic diseases.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  Time from randomization to disease recurrence or death of any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
Treatment-related adverse events assessed by CTCAE v4.0 | 3 years

IPD SHARING:
Plan to Share IPD: No
no plan to share data